CLINICAL TRIAL: NCT01088425
Title: Maternal Pregnancy and Neonatal Outcome After Assisted Reproduction. Comparison of Vitrification vs. Spontaneous Conception
Brief Title: Vitrification Versus Spontaneous Conception and Slow- Rate Freezing
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Daniel Alexander Beyer, Dr. D. A. Beyer, University of Luebeck
Other Study IDs: UKSH-HL-09-195; 09-195 (Registry Identifier: Ethik- Kommission zu Lübeck)
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Pregnancy
Keywords: vitrification; 2PN oocyte; maternal and infant health; embryo survival, clinical pregnancy rate; mode of delivery; injury during delivery; infant development; infant morbidity; slow- rate freezing
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Spontaneous: Mothers with children conceived after spontaneous cycle
  Interventions: Other: Observation
- Vitrificatíon: Mothers with children conceived after vitrification cycle
  Interventions: Other: Observation
- slow- rate freezing: Mothers with children conceived after slow- rate freezing cycle
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Alberta infant motor scale
  Griffiths test
  Kauffmann ABC

SUMMARY:
Great scientific effort has been made to improve practical as well as economical procedures of modern assisted reproduction.

In the last years a shift from the well established method of slow-rate freezing to vitrification of 2PN zygotes and embryos could be observed. Like any other method of cryopreservation, the outcome of vitrification will be affected by several factors related to technique itself, its practical management and patient characteristics.

The investigators want to investigate the influence of vitrification on the outcome of of 2PN oocytes, pregnancy and infant health.

A Comparison between a cohort of spontaneous conceived children and children of vitrified and slow- cooled 2PN oocytes is planned.

ELIGIBILITY:
Inclusion Criteria:

* cryopreservation (vitrification and slow- rate freezing) between 1998 - 2010
* Treatment in Lübeck University
* Delivery in Lübeck University
* Positive informed consent

Exclusion Criteria:

* Negative informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: tertiary university hospital
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maternal pregancy outcome | 7 years
  spontaneous or operative delivery, birth injuries, conjoined morbidity
embryo survival | 7 years
  embryo survival rate

SECONDARY OUTCOMES:
infant health | 7 years
  infant vital characteristics (APGAR, arterial cord ph), infant development: only develomental milestones: sitting, standing, walking infant morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Beyer, MD, Principal Investigator — Lübeck University
Locations (1):
- Schleswig- Holstein University, Campus Lübeck, Department of Reproductive Medicine, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Wennerholm UB, Soderstrom-Anttila V, Bergh C, Aittomaki K, Hazekamp J, Nygren KG, Selbing A, Loft A. Children born after cryopreservation of embryos or oocytes: a systematic review of outcome data. Hum Reprod. 2009 Sep;24(9):2158-72. doi: 10.1093/humrep/dep125. Epub 2009 May 20. PMID 19458318
- [Background] Kagawa N, Kuwayama M, Nakata K, Vajta G, Silber S, Manabe N, Kato O. Production of the first offspring from oocytes derived from fresh and cryopreserved pre-antral follicles of adult mice. Reprod Biomed Online. 2007 Jun;14(6):693-9. doi: 10.1016/s1472-6483(10)60670-0. PMID 17579980
- [Background] Noyes N, Porcu E, Borini A. Over 900 oocyte cryopreservation babies born with no apparent increase in congenital anomalies. Reprod Biomed Online. 2009 Jun;18(6):769-76. doi: 10.1016/s1472-6483(10)60025-9. PMID 19490780
- [Background] Noyes N, Knopman J, Labella P, McCaffrey C, Clark-Williams M, Grifo J. Oocyte cryopreservation outcomes including pre-cryopreservation and post-thaw meiotic spindle evaluation following slow cooling and vitrification of human oocytes. Fertil Steril. 2010 Nov;94(6):2078-82. doi: 10.1016/j.fertnstert.2010.01.019. Epub 2010 Feb 26. PMID 20188356
- [Background] Ubaldi F, Anniballo R, Romano S, Baroni E, Albricci L, Colamaria S, Capalbo A, Sapienza F, Vajta G, Rienzi L. Cumulative ongoing pregnancy rate achieved with oocyte vitrification and cleavage stage transfer without embryo selection in a standard infertility program. Hum Reprod. 2010 May;25(5):1199-205. doi: 10.1093/humrep/deq046. Epub 2010 Feb 25. PMID 20185513
- [Background] Al-Hasani S, Ozmen B, Koutlaki N, Schoepper B, Diedrich K, Schultze-Mosgau A. Three years of routine vitrification of human zygotes: is it still fair to advocate slow-rate freezing? Reprod Biomed Online. 2007 Mar;14(3):288-93. doi: 10.1016/s1472-6483(10)60869-3. PMID 17359578